CLINICAL TRIAL: NCT06849167
Title: A Single-Arm Phase II Clinical Trial of Immunotherapy Combined with Hypofractionated Concurrent Chemoradiotherapy Followed by Immunotherapy in Patients with Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Immunotherapy Combined with Hypofractionated Concurrent Chemoradiotherapy Followed by Immunotherapy in LA-NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Huiming Yu, Peking University Cancer Hospital & Institute (PekingUCHI), Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGH2024453
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Immunotherapy; Non-Small Cell Lung Cancer; hypofractionated radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hypofractionated group (Experimental): Immunotherapy combined with hypofractionated concurrent chemoradiotherapy followed by consolidation immunotherapy
  Interventions: Radiation: hypofractionated radiotherapy with immunotherapy

INTERVENTIONS:
Radiation: hypofractionated radiotherapy with immunotherapy — Immunotherapy combined with hypofractionated concurrent chemoradiotherapy followed by consolidation immunotherapy

SUMMARY:
Patients with locally advanced NSCLC (Non-Small Cell Lung Cancer) who have a PD-L1 TPS ≥ 20% will be included in this study. It aims to explore the efficacy and safety of immunotherapy combined with hypofractionated concurrent chemoradiotherapy, followed by consolidation immunotherapy.

Participants will undergo large fractionated radiotherapy with a total dose of 48Gy/16 fractions, 3Gy per fraction, 5 days a week. Participants will receive two cycles of concurrent platinum-based doublet chemotherapy and concurrent immunotherapy. Patients without progression will receive consolidation immunotherapy. The maximum duration of immunotherapy is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent before implementing any trial-related procedures.
2. Age ≥ 18 years and ≤ 70 years, male or female.
3. Histologically or cytologically confirmed inoperable locally advanced (IIB-IIIC) NSCLC (International Association for the Study of Lung Cancer and American Joint Committee on Cancer 8th edition TNM lung cancer staging);

   Notes:
   1. If EBUS/EUS or mediastinoscopy can safely obtain samples from the hilar or mediastinal lymph nodes, it is encouraged to obtain tissue for confirmation of involvement. When the lymph node boundary is clear and at least one lymph node has a short axis ≥ 2.0 cm, lymph node involvement can be determined by imaging (CT/MRI scan). For lymph nodes with a short axis < 2.0 cm, if pathologically confirmed, the patient can be included in the study. If the primary tumor is deemed unresectable and mediastinal lymph node metastasis does not affect the radiotherapy plan, the patient can be included.
   2. Determined and documented by a multidisciplinary tumor board or consultation with a thoracic surgeon: the patient has inoperable stage IIB-IIIC NSCLC.
4. No evidence of distant metastatic disease on diagnostic quality CT or MRI scans of the chest, abdomen, pelvis, and brain and/or whole-body fluorodeoxyglucose (FDG)-PET/CT, and classified as non-IV stage NSCLC (i.e., M0).

   Note: For pleural effusion present in both CT chest scan and frontal chest X-ray, a thoracentesis should be performed to confirm the pleural effusion is negative on cytology and is non-exudative. For patients who meet all other inclusion/exclusion criteria but are unable to undergo thoracentesis due to minimal pleural effusion, they may still be included in the study.
5. Provide a sufficient amount of quality-controlled tumor tissue or cell wax blocks for the pathology department of the study center to test PD-L1 expression using the 22C3 antibody, with a PD-L1 TPS ≥ 20%; or a pre-screening PD-L1 TPS ≥ 20% result (regardless of the antibody used, including 22C3, SP263, SP142).
6. At least one measurable lesion based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for use as a target lesion.
7. No prior treatment for advanced/metastatic NSCLC (chemotherapy, targeted therapy, immunotherapy, or radiotherapy). Patients who have previously received systemic induction or neoadjuvant therapy (chemotherapy, immunotherapy) for stage IIB-IIIC NSCLC and are about to receive curative concurrent chemoradiotherapy can be included in the study.
8. Patients who have previously received induction immunotherapy can be included, including the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or drugs targeting another co-stimulatory or inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137), immune LAG-3 inhibitors, and TIGIT monoclonal antibodies.
9. ECOG performance status of 0-1.
10. Life expectancy ≥ 6 months.
11. Adequate organ function, with the following laboratory parameters:
12. For women of childbearing potential, a negative urine or serum pregnancy test must be performed within 3 days prior to the first dose of study drug (Day 1 of Cycle 1). If the urine pregnancy test cannot be confirmed as negative, a serum pregnancy test is required. Non-childbearing potential women are defined as those who are at least 1 year post-menopausal, surgically sterilized, or have undergone a hysterectomy.
13. If there is a risk of pregnancy, all participants (regardless of sex) must use a contraceptive method with a failure rate of less than 1% during the entire treatment period and for 120 days after the last dose of the study drug (or 180 days after the last dose of chemotherapy).

Exclusion Criteria:

1. Pathologically diagnosed small cell lung cancer (SCLC), or mixed tumors containing small cell components.
2. Have undergone genetic testing prior to enrollment and known to have sensitive mutations in EGFR, ALK, or ROS-1 genes.
3. Subjects evaluated by the investigator with cavitary squamous carcinoma or imaging suggesting large vessel invasion/infiltration, or those with a history of active hemoptysis (coughing up at least 1/2 teaspoon of fresh blood) within 2 weeks prior to the first dose of the study drug.
4. In the planned radiotherapy regimen, the volume of normal lung tissue (total lung - GTV) receiving a total radiation dose >20Gy may exceed 34%.

   Have previously received any chest-directed radiotherapy (including esophagus, mediastinum, or breast cancer radiotherapy) before the first dose of the study drug.
5. Have undergone major surgery within 3 weeks prior to the first dose of the study drug (excluding surgeries for biopsy purposes or vascular access placement, but subjects must have fully recovered from treatment toxicities and/or complications).
6. Have been diagnosed with a malignancy other than NSCLC within 5 years prior to the first dose (excluding surgically cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or surgically resected carcinoma in situ).
7. Are currently participating in an interventional clinical trial or have received other investigational drugs or used investigational devices within 4 weeks prior to the first dose, or are expected to require any other form of anti-tumor treatment during the study.
8. Have received traditional Chinese medicine with anti-lung cancer indications or immune-modulating drugs (including thymosin, interferons, interleukins) as systemic treatment within 2 weeks prior to the first dose of the study drug.
9. Have had active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years prior to the first dose of the study drug. Alternative therapies (e.g., thyroid hormones, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatments.
10. Are receiving systemic glucocorticoid therapy (excluding nasal, inhaled, or other forms of local glucocorticoid therapy) or any other form of immunosuppressive therapy within 7 days before the first dose of the study drug.

    Note: Physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are allowed.
11. Specific to pemetrexed: If aspirin or other NSAIDs cannot be discontinued for at least 2 days before, during, and 2 days after pemetrexed administration (except when daily aspirin dose is ≤1.3g), or the patient cannot or refuses to take folic acid, vitamin B12, and dexamethasone.
12. Have known history of organ transplantation (excluding corneal transplants) or allogeneic hematopoietic stem cell transplantation.
13. Have known allergies to any of the active ingredients or excipients of the study drugs, including PD-1/PD-L1 monoclonal antibodies, pemetrexed, injectable albumin-bound paclitaxel, paclitaxel, carboplatin, cisplatin, etc.
14. Have a history of bleeding tendencies (e.g., active gastrointestinal ulcers) or are receiving anticoagulants or vitamin K antagonists such as warfarin, heparin, or its analogs.

    Note: Small-dose warfarin (≤1mg/day), low-dose heparin (≤12,000 U/day), or low-dose aspirin (≤100mg/day) may be used for prophylactic purposes if the international normalized ratio (INR) is ≤1.5.
15. Have experienced severe arterial/venous thromboembolic events (e.g., cerebrovascular accident, including transient ischemic attacks, deep vein thrombosis, or pulmonary embolism) within 6 months prior to the first dose.
16. Have not fully recovered from any toxicity and/or complications from previous interventions (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss).
17. Have a known history of human immunodeficiency virus (HIV) infection (i.e., HIV1/2 antibody positive).
18. Have untreated active hepatitis B (defined as HBsAg positive and HBV-DNA levels exceeding the upper normal limit at the local center's laboratory).

    Note: The following hepatitis B patients may be included:

    HBV viral load <1000 copies/ml (200 IU/ml) before the first dose, provided they receive anti-HBV treatment throughout the study period to prevent viral reactivation.

    Subjects who are anti-HBc (+), HBsAg (-), anti-HBs (-), and have HBV viral load (-) do not need prophylactic anti-HBV treatment but should be closely monitored for viral reactivation.
19. Have active HCV infection (HCV antibody positive with HCV-RNA levels above the detection threshold).
20. Have received a live vaccine within 30 days prior to the first dose of the study drug (Day 1, Cycle 1).

    Note: Inactivated seasonal influenza vaccines and COVID-19 vaccines for prevention are allowed within 30 days prior to the first dose, but live attenuated influenza vaccines administered intranasally are not permitted.
21. Are pregnant or breastfeeding women.
22. Have any severe or uncontrolled systemic diseases
23. Any other medical history or evidence of disease, treatment, or abnormal laboratory findings that may interfere with the study results or hinder participation, or any other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 3 years
  From subject enrollment to the first recorded disease progression or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
ORR | through study completion, an average of 3 years
  The proportion of subjects achieving complete response (CR) or partial response (PR) as their best overall response following treatment initiation, relative to the total number of subjects.
DCR | through study completion, an average of 3 years
  The proportion of subjects achieving complete response (CR), partial response (PR), or stable disease (SD) as their best overall response following treatment initiation, relative to the total number of subjects.
DOR | through study completion, an average of 3 years
  Time interval from the first documented evidence of response (CR or PR) to disease progression or death (whichever occurs first).
OS | through study completion, an average of 3 years
  Time from subject enrollment to death from any cause.
HRQoL Assessment: | through study completion, an average of 3 years
  The "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 items" (EORTC QLQ-C30) will be used to evaluate subjects' global health status.
Safety Evaluation | through study completion, an average of 3 years
  Adverse events (AEs) occurring during the study and follow-up period will be graded for severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0). Safety evaluation metrics include:
  Incidence, severity, and relationship to study treatment of all adverse events (AEs), treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and immune-related adverse events (irAEs); Number and proportion of subjects discontinuing treatment due to the above adverse events;
Economic Evaluation | through study completion, an average of 3 years
  Cost-effectiveness of medical interventions will be assessed using metrics such as the Incremental Cost-Effectiveness Ratio (ICER) and Quality-Adjusted Life Years (QALYs).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China